CLINICAL TRIAL: NCT01839474
Title: Clinical Trial Evaluating the Difference in Mortality Rates in Children in Ghana Receiving CPAP Versus Those Who Do Not
Brief Title: CPAP Survival Study in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Kwame Nkrumah University of Science and Technology (Other)
Responsible Party: Principal Investigator, Rachel Moresky, Assistant Clinical Professor of Population & Family Health and Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ7954; GENERAL ELECTRIC FOUNDATION (Other Grant/Funding Number: PT-AABF5157)
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Pneumonia; Acute Respiratory Infection
Keywords: Continuous Positive Airway Pressure; Controlled trial; Pneumonia; Children
MeSH Terms: conditions — Pneumonia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP (Experimental): Children will be placed on nasal CPAP until they have an age appropriate respiratory rate and receive standard medical therapy.
  Interventions: Device: CPAP
- Control (No Intervention): Children will receive standard medical therapy.

INTERVENTIONS:
Device: CPAP — Appropriately sized nasal prongs will be selected for the patient, gently applied ensuring a tight seal, and securely fastened. The CPAP machine will be turned on to deliver a pressure of 5 cm H2O in the inspiratory limb of the system. Patients will be allowed to be in the position of most comfort, preferably with mouth closed to maintain pressure in the circuit.
  Other Names: Continuous Positive Airway Pressure
  Arms: CPAP

SUMMARY:
The purpose of this study is to determine if the use of a continuous positive airway pressure (CPAP) machine (a device that blows air into the lungs) decreases the chance of a child dying from difficulty breathing.

DETAILED DESCRIPTION:
Acute respiratory infections, malaria, and sepsis remain leading causes of death in children throughout the world.These conditions may lead to respiratory distress and eventually failure if not adequately managed. In developing countries with limited resources, advanced airway management and support can be challenging and needs to be approached in a different manner than is done in developed nations. For example, the use of invasive mechanical ventilation for respiratory distress is not an option in many resource-limited countries due to the lack of available technology, infrastructure, and trained personnel. Other alternatives should be utilized in order to support children with reversible conditions during their acute respiratory distress stage. One such alternative is non-invasive positive pressure.

Prior research demonstrated that nasal bubble CPAP can be successfully introduced and utilized in a developing country's emergency ward. Nurses in four Ghanaian district hospital emergency wards (Kintampo, Mampong,Nkoranza, and Wenchi) were able to safely apply CPAP and monitor the patient's response. The investigators demonstrated that patients receiving CPAP had a significant decrease in respiratory rate compared with those that did not with a mean difference of 14 breaths per minute. There were no major side effects associated with the use of CPAP. Now that CPAP has demonstrated to decrease respiratory rate in a non-specific disease population presenting with respiratory distress it is important to determine if it also improves survival. Therefore, the purpose of the study is to determine if the use of CPAP in children 1 month to 5 years of age with respiratory distress decreases mortality.

ELIGIBILITY:
Inclusion Criteria:

* One month to five years of age
* Respiratory rate (RR) greater than 50 breaths per minute in three months to one year of age, and greater than 40 breaths per minute in one to five years of age
* Presence of sub costal, intercostal, supraclavicular retractions or nasal flaring

Exclusion Criteria:

* Age less than one month or older than five years
* Skin breakdown around nose/mouth or facial trauma
* Unable to protect airway
* Uncontrollable emesis
* Unresponsiveness
* poor respiratory effort requiring positive pressure ventilation or invasive mechanical ventilation for respiratory failure
* known or suspected pneumothorax

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2200 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 2 weeks
  The primary outcome will be 2 week mortality rate in children receiving CPAP and standard therapy compared with children receiving standard therapy alone.

SECONDARY OUTCOMES:
Respiratory rate | 24 hours
  To measure change in respiratory rates between children receiving CPAP compared to those who do not for 24 hours.

OTHER OUTCOMES:
Evidence of viral respiratory infection | baseline (at time of enrolment)
  To determine the etiology of respiratory distress. We will test nasopharyngeal swabs for common pediatric viruses.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel T Moresky, MD, MPH, Principal Investigator — Columbia University
Locations (2):
- Ghana (2):
  - Mampong District Hospital, Mampong, Ashanti Region
  - Kintampo District Hospital, Kintampo, Brong Ahafo

REFERENCES:
- [Derived] Wilson PT, Baiden F, Brooks JC, Morris MC, Giessler K, Punguyire D, Apio G, Agyeman-Ampromfi A, Lopez-Pintado S, Sylverken J, Nyarko-Jectey K, Tagbor H, Moresky RT. Continuous positive airway pressure for children with undifferentiated respiratory distress in Ghana: an open-label, cluster, crossover trial. Lancet Glob Health. 2017 Jun;5(6):e615-e623. doi: 10.1016/S2214-109X(17)30145-6. PMID 28495265